CLINICAL TRIAL: NCT05049876
Title: Prevalence of Renal Disease in Children With Celiac Disease
Acronym: COELIGAN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200251; IDRCB: 2020-A00316-33 (Registry Identifier: ANSM)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-07

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: urine sample taken during consultations — urine sample taken during consultations

SUMMARY:
To assess the prevalence of renal disease in a pediatric population of patients with celiac disease by looking for the presence of hematuria and/or proteinuria.

DETAILED DESCRIPTION:
In this study the investigators seek to quantify the prevalence of urine sediment abnormalities in children with celiac disease to assess whether there is value in screening for renal disease in this population. Celiac disease (CD) is frequently accompanied by a variety of extra-digestive manifestations, making it a systemic disease rather than a disease limited to the gastrointestinal tract. CD belongs to the group of autoimmune diseases, a significantly increased prevalence of other autoimmune diseases (AD) has been reported in individuals with CD and their first-degree relatives, and a significantly increased prevalence of CD has been documented in individuals with other AD. The association between CD and other ADs may be explained by a shared pathogenic basis, involving genetic susceptibility as in type 1 diabetes (T1D), similar environmental triggers, increased intestinal permeability, and possibly by undiscovered mechanisms. Many of the extraintestinal manifestations of CD involve the kidney. Urolithiasis and crystal-induced renal disease, nephrogenic ascites, increased risk of end-stage renal disease, and membranoproliferative glomerulonephritis type 1 are associated with CD. However, little is known about the risk of kidney disease in individuals with CD, and it would be interesting to assess the prevalence of urine sediment abnormalities in a pediatric population at diagnosis and during follow-up. No previous studies have examined the risk of renal disease, and there are currently no recommendations for screening for renal involvement in patients with CD.

One of the renal conditions that particularly attracts our attention is IgA nephropathy (NIgA). First, studies suggest a common pathogenic basis between this nephropathy and CD and second, it is one of the most common primary glomerulonephritis in children and adolescents worldwide. NIgA usually progresses to end-stage renal disease (ESRD) within 20 years; the median age of patients starting dialysis ranges from 40 to 50 years. Cohort studies with extensive follow-up show that 10-13% of children eventually reach ESRD within 10 years and 20-30% within 20 years. In more than half of cases, NIgA is asymptomatic (microscopic hematuria) and is diagnosed after an incidental finding of hypertension, subnormal glomerular filtration rate, hematuria, and/or proteinuria in children and adults. Renin-angiotensin system inhibitors have shown effective results in reducing the progression of kidney damage in young NigA patients with moderate proteinuria.

In view of its potential severity, the arguments in favor of its association with CD, its generally asymptomatic clinical presentation, and the usefulness of its early detection, it seems interesting to us to evaluate the prevalence of urinary abnormalities characteristic of NigA in children with celiac disease. The results of this study could have an impact on the prevention of renal disease in patients with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* children with Celiac Disease

Exclusion Criteria:

-

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children with Celiac Disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
urine sediment abnormalities (proteinuria , creatininuria) | 1 day
  measurement of proteinuria, creatininuria and urine cytology Hematuria is defined by a number of red blood cells in the urine greater than or equal to 10,000 / ml. This will be carried out by counting red blood cells by an automatic device.
  The search for proteinuria will be carried out on a urination by an automatic device. Proteinuria is considered positive when the urine protein / creatinine ratio is 0.03 g / mmol. In case of positive proteinuria we will measure the microalbuminuria on the same sample.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Baylet Fernandez, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No